CLINICAL TRIAL: NCT05594901
Title: Impact of a Risk Stratification Tool on the Outcome of Liver Transplant Recipients Colonized With Carbapenem Resistant Enterobacteriaceae: an Observational Study
Status: Active, not recruiting | Type: Observational
Sponsor: University of Bologna (Other)
Collaborators: The Mediterranean Institute for Transplantation and Advanced Specialized Therapies (Other); ASST-Sette Laghi Università degli Studi dell'Insubria Varese (Unknown); Università degli Studi di Padova Unit Multivisceral Transplant Unit Padova (Unknown); Università degli Studi di Verona - Gastroenterologia Verona (Unknown); Hospital General Universitario Gregorio Marañon (Other); Hospital das Clinicas da Faculdade de Medicina da Universidade de São Paulo São Paulo (Unknown)
Responsible Party: Principal Investigator, Maddalena Giannella, Associate Professor, University of Bologna
Other Study IDs: CRECOOLT 3.0
Record Dates: First submitted 2022-10-12; First posted 2022-10-26 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Liver Transplantation; Carbapenem-Resistant Enterobacteriaceae Colonization

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Retrospective Cohort
- Prospective Cohort
  Interventions: Other: Application of a prognostic score

INTERVENTIONS:
Other: Application of a prognostic score — The CRECOOLT score, for the prospective cohort, will be systematically calculated once week, or at the occurrence of complications, until 60 days after OLT. The therapeutic management of all patients, during both retrospective and prospective periods, will be established by the attending physicians according with routine practice and not dictated by study protocol.
  Groups: Prospective Cohort

SUMMARY:
Although CRE infection after OLT have a dramatic impact on patient survival and several implementations have been proposed (i.e. preventive strategies or targeted surgical prophylaxis), a standardized approach in colonized patients is still missing. The investigators recently developed and internally validated a bed-side score to stratify the risk of CRE infection in OLT recipients colonized by CRE. The goal of this pre/post observational study is to investigate the impact on all-cause 90-day mortality in OLT recipients colonized with CRE using such score (CRECOOLT score) for the systematic evaluation of CRE infection risk.

The secondary objectives are:

* To analyse days of therapy with anti-CRE antibiotic regimens in patients with and without systematic evaluation of CRE infection risk, according to clinical practices.
* To evaluate rates of documented CRE infections and their relapses with selection of further resistance in patients with and without systematic evaluation of CRE infection risk.
* To evaluate the length of hospital, ICU stay and rates of hospital readmission in patients with and without systematic evaluation of CRE infection risk.

DETAILED DESCRIPTION:
Patients undergoing orthotopic liver transplantation (OLT) are more susceptible to acquire colonization with multidrug resistant Gram-negative bacteria, in particular with carbapenem resistant Enterobacterales (CRE), than non-solid organ transplant (SOT) recipients or patients with other types of SOT. CRE colonization, either acquired before either emerged after OLT, has been associated with highest risk of developing CRE infection after OLT with a dramatic impact on patient survival. For these reasons, along with the improvement of infection control and antimicrobial stewardship policies, preventive strategies targeted to patients colonized with CRE have been suggested. However, several uncertainties have to be considered concerning the optimal timing for intervention, the correct patient stratification, and the choice of drugs. Regarding the timing for intervention, surgical prophylaxis is regarded as an option. However, it should be considered that of the overall burden of CRE carriage in OLT recipients, pre-transplant acquisition accounted for lower than one third of isolations in a large multicenter retrospective study. Furthermore, even when CRE carriage is present at transplantation, the colonization status is frequently recognized in the immediate post-operative period by results of rectal swabs done at surgery. Finally, current data about the efficacy of targeted prophylaxis in patients colonized with CRE are very limited and showed controversial results. Thus, in the majority of cases the unique window for preventive strategies is represented by the post-transplant course. This requires an active screening policy as well as the possibility of stratifying colonized patients according to their risk of developing CRE infection, and eventually to die, in order to target specific interventions in those patients who could most benefit, and to optimize essential resources as the new drugs. Indeed, since the availability of new drugs such as ceftazidime/avibactam, meropenem/vaborbactam and cefiderocol, the therapeutic management and outcome of patients colonized and/or infected with CRE has changed in both general population and SOT recipients. New drugs are associated with higher rates of clinical cure and patient survival, as well as with lower toxicity, compared with old regimens. However, rates of microbiological failure around 10%, consisting in persistent positive cultures or relapsing infections associated with development of further resistance, have been reported raising concerns about the need of optimizing the use of new drugs to avoid the loss of their efficacy.

To this end, the investigators have recently carried out a large multicenter observational study aimed at building a prediction model to stratify patients according to their risk of developing CRE infection after OLT. The study cohort consisted of 800 OLT recipients colonized with CRE, 25% were colonized at OLT, and 75% acquired colonization within two weeks after OLT. Infection rate was of 30% and was similar between the two groups as well as the infection severity. All-cause 6-month mortality rate among patients who developed CRE infection was 58% vs. 20% among carries who did not develop infection (p<0.001). Almost all infections occurred within 60 days after transplant. Thus, the investigators derived, and internally validated, a prediction tool able to stratify the risk of CRE infection at 30 and 60 days after OLT (CRECOOLT score) based on six variables easily to monitor such as CRE colonization detected in the 60 days prior to transplant, CRE colonization detected post-transplant, multisite colonization, need of prolonged (≥48 hours) mechanical ventilation, acute renal failure, and reintervention. The calculated cumulative incidence of CRE infection and nomogram-derived prediction for a low-risk and a high-risk patient were made available as app to be used bed-side. The investigators explored the potential clinical utility of our model using a decision-curve analysis to examine the "net benefit" of applying the prediction model across a range of CRE infection threshold probabilities. A theoretical risk-model guided strategy (i.e. empiric administration of CRE-active antibiotics) was compared against two default strategies- "treat all" and "treat none" suggesting that the model-directed intervention would show net benefit over default strategies when the overall CRE infection risk exceeded 10%.

Finally, the investigators have explored the risk of death using the same variables included in the CRECOOLT score by a multi-state model obtaining three risk groups: low, intermedium and high. The investigators have then estimated the potential impact of using ceftazidime-avibactam in each of such groups finding a significant protective role (HR 0.32) only in patients with intermedium or high risk of dying.

ELIGIBILITY:
Inclusion Criteria:

* Signature of the informed consent
* Age ≥ 18 years
* CRE colonization within 60 days prior to or after transplantation

Exclusion Criteria:

* Patients receiving targeted antibiotic prophylaxis (against CRE) for a period longer than 48 hours
* Patients receiving graft from a donor with cultures yielding a carbapenem-resistant Gram negative bacteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: OLT recipients colonized by CRE
Sampling Method: Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
The primary objective is to investigate the impact on all-cause 90-day mortality in OLT recipients colonized with CRE using the CRECOOLT score for the systematic evaluation of CRE infection risk. | 24 months

SECONDARY OUTCOMES:
To analyse days of therapy with anti-CRE antibiotic regimens in patients with and without systematic evaluation of CRE infection risk, according to clinical practices. | 24 months
To evaluate rates of documented CRE infections and their relapses. | 24 months
To evaluate the length of hospital and ICU stay (days) in patients with and without systematic evaluation of CRE infection risk. | 24 months
To evaluate selection of further resistance in patients with documented CRE infection relapse with and without systematic evaluation of CRE infection risk. | 24 months
To evaluate rates of hospital readmission in patients with and without systematic evaluation of CRE infection risk. | 24 months

CONTACTS AND LOCATIONS:
Locations (6):
- Hospital das Clinicas da Faculdade de Medicina da Universidade de São Paulo, São Paulo, Brazil
- Italy (4):
  - Università degli Studi di Padova - Unit Multivisceral Transplant Unit, Padua
  - Irccs Ismett, Palermo
  - ASST-Sette Laghi Università degli Studi dell'Insubria, Varese
  - Università degli Studi di Verona - Gastroenterologia, Verona
- Hospital General Universitario Gregorio Maranon, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-08-31): https://cdn.clinicaltrials.gov/large-docs/01/NCT05594901/Prot_SAP_000.pdf